CLINICAL TRIAL: NCT05186194
Title: The Effect of Vitamin D and Calcium Supplementation on the Prevention of Stress Fractures in Chinese Recruits.
Brief Title: The Effect of Vitamin D and Calcium Supplementation on the Prevention of Stress Fractures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20212116-F-2
Record Dates: First submitted 2021-12-08; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Stress Fracture; Vitamin d
MeSH Terms: conditions — Fractures, Stress | interventions — Vitamin D; Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Treatment) Group (Experimental): Oral vitamin D1000IU, 1/day, calcium 1200mg, 1/day, for 8 weeks.
  Interventions: Drug: Vitamin D, Calcium
- Control Group (Placebo Comparator): Oral placebo, for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D, Calcium — Vitamin D, calcium are available in tablets. During the 8 weeks of training, subjects were asked to take supplement tablets per day after dinner.
  Arms: Experimental (Treatment) Group
Drug: Placebo — Placebo
  Arms: Control Group

SUMMARY:
The main objective of this study is to find whether supplemental vitamin d and calcium can reduce the incidence of stress fractures in recruits. These high-risk recruits undergo intensive training which elevated bone turnover, which requires adequate level of vitamin D and calcium in order to support bone health. It is hypothesized that supplemental vitamin d and calcium will decrease the occurrence of stress fractures.

ELIGIBILITY:
Inclusion Criteria:

* Recruits newly enlisted at a training base in September 2021.
* Agree to accept relevant inspections and serological research, and sign an informed consent form.

Exclusion Criteria:

* Suffer from diabetes, osteomyelitis and other diseases.
* Suffer from claustrophobia and other MRI examination contraindications.
* Long-term use of glucocorticoids, non-steroidal anti-inflammatory drugs or calcium, vitamin D.
* A history of kidney disease.
* Allergic to any ingredient of the medicine.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Stress fracture | 3 months after the start of the basic military training.
  Stress fractures were recorded when recruits reported to the clinic with suspected symptoms. All stress fractures were confirmed with radiography or Magnetic Resonance Imaging(MRI). Each subject with a stress fracture was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Xijing Hospital, The Air Force Medical University, Xi’an, Shanxi, China